CLINICAL TRIAL: NCT05105880
Title: The Effectiveness of Cardio-auscultation and Pulse Oximetry Combined Screening of Congenital Heart Disease in Newborns
Brief Title: Auscultation and Pulse Oximetry Combined Screening of Neonatal Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Women and Children's Hospital of Linyi City (Other)
Responsible Party: Sponsor
Other Study IDs: CHDScreening
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Congenital Heart Disease
Keywords: Pulse oximetry; Auscultation; Congenital Heart Disease; Screening
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conducted this retrospective study in a large single center with an annual birth of more than 20,000 newborns, from January 1, 2018 to December 31, 2019, to confirm the applicability and accuracy of pulse oximetry (POX) combined cardio-auscultation to screen congenital heart disease for neonates.

DETAILED DESCRIPTION:
All consecutive newborn babies were eligible, irrespective of gestational age, NICU admission, symptom presence or prenatal diagnosis.

This study was approved by institutional ethical review board of Linyi Maternal and Child Healthcare Hospital. Spoken informed consent was obtained from the participating babies' parents.

Physicians from departments of neonatal medicine and developmental medicine undertake auscultation screening. When abnormal murmur occurred, an echocardiography would be requested to confirm if the newborn has CHD or not.

Physicians from obstetrics department and nursing staff from neonatal department undertake POX measurement. If a positive POX occurred, an echocardiography would be requested to confirm if the newborn has CHD or not.

Physicians from department of ultrasonography undertake echocardiography confirmation for newborns deemed positive by auscultation or POX.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive newborn babies delivered in the study center were eligible, irrespective of gestational age, NICU admission, symptom presence or prenatal diagnosis.

Exclusion Criteria:

* None.

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population focus on the neonates delivered in the two campuses of the study center which is the largest maternal facility in a municipality of 11 million population.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Severe congenital heart disease | The first 24 hours after birth.
  Patients who present as severely ill in the newborn period or early infancy, including those with cyanotic heart disease and acyanotic lesions like AVSD, large VSD, large PDA, critical or severe AS, severe PS, critical coarc.

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Children's Hospital of Linyi City, Linyi, Shandong Provicne, China

IPD SHARING:
Plan to Share IPD: Undecided